CLINICAL TRIAL: NCT00000936
Title: Controlled Trial of Induction Therapy in Renal Transplantation
Brief Title: A Study To Test An Anti-Rejection Therapy After Kidney Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT IN01/OLN-359
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Induction (Experimental): subjects receiving hOKT3 induction therapy
  Interventions: Drug: hOKT3; Drug: Oral Cyclosporine
- Induction Free Therapy (Active Comparator): Patients not receiving induction therapy
  Interventions: Drug: Oral Cyclosporine; Drug: IV Cyclosporine

INTERVENTIONS:
Drug: hOKT3 — Administered both during and after transplantation in IV form. Dosage determined by individual weight and given for a maximum of 14 days.
  Arms: Induction
Drug: Oral Cyclosporine — Administered orally as either sandimmune or neoral at a dose determined by weight. Patients 6 years of age and older begin at a dose of 15 mg/kg/day and patients under 6 years of age receive 500 mg/m2/day, for the duration of the study.
Drug: IV Cyclosporine — Administered intravenously (IV) both during and after transplantation at a dosage determined by individual age.
  Arms: Induction Free Therapy

SUMMARY:
Kidney transplantation is often successful. However, despite aggressive anti-rejection drug therapy, some patients will reject their new kidney. This study is designed to test two anti-rejection approaches. Two medications in this study are currently used in children, but there is no information regarding which drug is safer or more effective.

Survival rates in renal transplantation are unacceptably low. Therefore, there is a need for an improved post-transplant treatment, such as the induction therapy used in this study.

DETAILED DESCRIPTION:
Renal transplantation is recognized as the treatment of choice for children with chronic renal failure. However, patient and graft survival rates in young children are unacceptably low. In preliminary studies, OKT3 (a monoclonal antibody) induction therapy received post transplant has been more successful than standard immunosuppression alone in improving graft survival. This study is designed to assess the impact of induction therapy on graft survival in pediatric kidney transplant patients.

Patients are assigned to OKT3 induction or no induction in a 1:1 ratio. Randomization to oral cyclosporine of either Sandimmune or Neoral is also done in a 1:1 ratio. Group 1 receives OKT3 intraoperatively followed by Neoral. Group 2 receives OKT3 intraoperatively followed by Sandimmune. OKT3 is administered at 2.5 mg (if weight less than 30 kg) or 5 mg (if weight above 30 kg) per day for a maximum of 14 days. Group 3 receives IV cyclosporine followed by Neoral. Group 4 receives IV cyclosporine followed by Sandimmune. Oral cyclosporine is administered in a masked preparation. The dose for Sandimmune and Neoral is the same; patients 6 years of age and older begin at a dose of 15 mg/kg/day and patients under 6 years of age receive 500 mg/m2/day. Patients will receive concomitant medications including steroids (IV and po), Nifedipine, anti-CMV therapy, Bactrim, Azathioprine or Mycophenolate Mofetil. Kidney function, incidence of viral infection, graft survival, and incidence of malignancy will be measured to assess the role of OKT3 induction and the role of rejection in graft failure. Graft function will be evaluated at 1-, 2-, and 4-year intervals.

ELIGIBILITY:
Inclusion Criteria

Children and young adults may be eligible for this study if they:

* Are not yet 21 years of age.
* Are receiving their first or second transplant.
* Are not pregnant.
* Agree to practice sexual abstinence or agree to use an effective
* method of birth control/contraception during the study and
* for 1 year after.

Exclusion Criteria

Children and young adults will not be eligible for this study if they:

* Are recipients of multiple organs other than kidneys.
* Are recipients of three or more transplants.
* Are HIV positive.
* Are Hepatitis B surface antigen positive.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 292 (Actual)
Dates: Start 1999-11; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
To determine one-year graft function, as measured by graft survival and serum creatinine of children undergoing OKT3 induction versus no induction | At 1 year
To compare the efficacy of Sandimmune and Neoral with respect to graft function | Throughout study

SECONDARY OUTCOMES:
Two and four-year graft functions | At 2 and 4 years
Safety with respect to viral infections and malignancies in children undergoing a renal transplant | Throughout study
Frequency and severity of rejection episodes | Throughout study
Time to first rejection | Throughout study
Length and frequency of hospitalization | Throughout study
Nature of acute cellular rejection at a molecular level | Throughout study
Nature of "heightened immune response" of younger children by studying gene expression in surveillance biopsies | Throughout study
Correlate intragraft events during rejection with cytokine profile in the peripheral blood | Throughout study

CONTACTS AND LOCATIONS:
Locations (1):
- Ilene Blechman-Krom, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- See also: The National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY354 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY354 — ImmPort study identifier is SDY354.
- Available data/document: Study Protocol: SDY354 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY354 — ImmPort study identifier is SDY354.
- Available data/document: Study summary, -design, -demographics, -lab tests, -study files: SDY354 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY354 — ImmPort study identifier is SDY354.